CLINICAL TRIAL: NCT01788189
Title: Lenalidomide in Conjunction With Methotrexate, Leucovorin, Cytarabine and Rituximab for the Treatment of Relapsed or Refractory CD20-positive Aggressive Lymphomas: an Open-label, Multicenter Phase I/II Trial
Brief Title: Lenalidomide, MTX, Ara-C and Rituximab in Relapsed Aggressive B-cell Lymphomas
Acronym: LeMLAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Ulrich Duehrsen, Prof. Dr. med., University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No. 2012-001891-13
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: B-cell Lymphoma
Keywords: Lymphoma; CD20; Relapse; Lenalidomide
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental): The LeMLAR protocol:
  Lenalidomide 25 mg p.o., days 1 - 21; Methotrexate 30 - 60 - 90 - 120 - 150 mg/m² i.v. bolus, days 1, 8, 15; Leucovorin 4 x 45 mg p.o. (every 6 hrs), days 2, 9, 16; Cytarabine (Ara-C) 75 - 150 - 225 - 300 - 375 mg/m² i.v. bolus, days 1, 8, 15; Rituximab 375 mg/m² i.v. infusion, day 1.
  28-day cycles, maximum 6 cycles, definition of dose-limiting toxicity in cycles 1 and 2, intra-patient dose escalation after cycles 2 and 4 in case of absence of dose-limiting toxicity in previous cycles
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide

SUMMARY:
Multicenter prospective open-label non-randomised phase I/II study in patients with relapsed or refractory CD20-positive aggressive lymphomas

Phase I:

Dose escalation of methotrexate and cytarabine (days 1, 8 and 15 of each 28-day cycle) in a 3 + 3 design with fixed doses of lenalidomide (days 1 - 21) and rituximab (day 1), maximum 6 cycles

Phase II:

Treatment of 20 patients at maximum tolerated doses of phase I

DETAILED DESCRIPTION:
Phase I

The goal of the phase I part of the study is to determine the maximum tolerated doses of methotrexate and cytarabine able to be combined with once-per-cycle rituximab and full-dose 3-weeks-on/1-week-off lenalidomide in 28-day treatment cycles. Methotrexate and cytarabine will be given three times per cycle, preferably on days 1, 8 and 15. If short-term toxicity precludes once-per-week dosing, treatment may be delayed by a maximum of 3 days, e.g. the second injection of methotrexate and cytarabine may be delayed until day 11 and the third injection until day 21. The doses of methotrexate and cytarabine will be adjusted to permit administration of three doses per cycle without the need to postpone the subsequent treatment cycle by more than 7 days.

Dose limiting toxicity will be determined by increasing the doses of methotrexate and cytarabine in sequential patient cohorts in a 3 + 3 design. Because tolerance to lenalidomide and cytotoxic agents are likely to decrease with increasing numbers of treatment cycles, evaluation of dose-limiting toxicity will be confined to the first two cycles. The requirement for dose reductions in subsequent treatment cycles will not be rated as dose-limiting toxicity.

If no dose-limiting toxicity is observed in 3 patients treated at the same dose level, the next 3 patients will be treated at the next higher dose level. If a single patient experiences dose-limiting toxicity, another 3 patients will be treated at the same dose level. If no more than one dose-limiting toxicity is observed in 6 patients treated at that level, the next 3 patients will be treated at the subsequent dose level. If two or more of 3 - 6 patients treated at the same level experience dose-limiting toxicity, dose escalation will be stopped. The dose level below the level where dose-limiting toxicity was observed defines the maximum tolerated dose.

The dose level below the level where dose-limiting toxicity is observed defines the maximum tolerated doses of methotrexate and cytarabine. However, if, at a lenalidomide dose of 25 mg, methotrexate and cytarabine cannot be escalated beyond the first dose level, the lenalidomide dose will be reduced to 20 mg, and the methotrexate/cytarabine dose level producing dose-limiting toxicity will be repeated at a lenalidomide dose of 20 mg. If, at a lenalidomide dose of 20 mg, methotrexate and cytarabine cannot be escalated beyond the first dose level, the lenalidomide dose will be reduced to 15 mg, and the methotrexate/cytarabine dose level producing dose-limiting toxicity will be repeated with a lenalidomide dose of 15 mg. If, at a lenalidomide dose of 15 mg, methotrexate and cytarabine cannot be escalated beyond the first dose level, dose limiting toxicity is reached and the maximum tolerated dose is the highest dose of lenalidomide able to be combined with the first dose level of methotrexate and cytarabine in a 3 + 3 phase I design.

The toxicity profiles of methotrexate (mucositis, hepatotoxicity) and cytarabine (hematotoxicity, hepatotoxicity) differ. In order to determine the maximum tolerated dose of each compound, further dose escalation of one or other drug may be required after the maximum tolerated dose of the methotrexate/cytarabine combination (as defined in dose levels 1 - 5, see below) has been determined. If dose-limiting hematotoxicity occurs without concomitant dose-limiting mucositis or hepatotoxicity, the dose of methotrexate may be escalated without concomitant increase of the cytarabine dose. Conversely, if severe mucositis occurs without concomitant dose-limiting hematotoxicity or hepatotoxicity, the dose of cytarabine may be escalated without concomitant increase of the methotrexate dose. Dose modifications of individual drugs will be made by the coordinating principal investigator according to the observed toxicities using the levels defined for the methotrexate/cytarabine combination.

Toxicities observed during the first two treatment cycles will be reported to the trial office within 7 days after their occurrence (in case of serious adverse events within 24 hours). Based on the predefined criteria listed below the coordinating principal investigator and the trial coordinator will decide whether or not a toxicity fulfils the requirements of a dose-limiting toxicity. After inclusion of up to 6 patients on the same dose level the coordinating principal investigator and the trial coordinator will decide according to the principles outlined in this protocol whether it is safe to move on to the next dose level. If rating a toxicity as dose-limiting is equivocal and/or no agreement is obtained between the coordinating principal investigator and the trial coordinator, the principal investigators of all participating trial sites will be included in the decision making process. Stepping-up to the next dose level will require more votes to be in favor of than against dose escalation.

Dose-limiting toxicities are:

* any of the following on the day of methotrexate/cytarabine injection (day 8 + ≤ 3 days / day 15 + ≤ 6 days of the first or second treatment cycle; day 1 of the second or third cycle which is equivalent to day 29 + ≤ 7 days of the previous cycle): neutrophils < 500/µl, platelets < 25.000/µl, creatinine clearance < 60 ml/min, bilirubin ≥ 3,0 mg/dl, serum AST/GOT or ALT/GPT ≥ 6 x upper limit of normal, mucositis grade 3 or 4
* requirement for dose reduction of methotrexate/cytarabine in the first or second treatment cycle
* fewer than 21 days of lenalidomide in the first or second treatment cycle
* toxicity-related delay of second or third treatment cycle by more than 7 days
* any other toxicity preventing continuation of therapy according to protocol in the first or second treatment cycle (except allergic reactions)

Depending on previous treatment history patients will vary in their tolerance to the LeMLAR regimen. To provide maximum therapeutic benefit, the doses of methotrexate and cytarabine will be escalated within individual patients after cycles 2 and 4 as detailed below provided no dose limiting toxicities occurred in previous treatment cycles. Dose escalation in cycles 3 to 6 in individual patients will not be used to determine dose-limiting toxicity. This will only be done in cycles 1 and 2.

Patients should receive 6 treatment cycles unless tumor progression, unacceptable toxicity or treatment intolerance occurs. Treatment intolerance includes physician or patient preference to discontinue or change treatment in a manner not compatible with the protocol. If treatment according to the LeMLAR protocol is prematurely stopped, its result must be documented by the procedures outlined in the protocol.

Definition of dose levels of methotrexate and cytarabine (cohorts of 3 - 6 patients):

Level 1

Cycles 1 - 2: methotrexate 30 mg/m², cytarabine 75 mg/m²; cycles 3 - 4: if no dose-limiting toxicity occurs in cycles 1 and 2: methotrexate 60 mg/m², cytarabine 150 mg/m²; cycles 5 - 6: if no dose-limiting toxicity occurs in cycles 3 and 4: methotrexate 90 mg/m², cytarabine 225 mg/m²

Level 2

Cycles 1 - 2: methotrexate 60 mg/m², cytarabine 150 mg/m²; cycles 3 - 4: if no dose-limiting toxicity occurs in cycles 1 and 2: methotrexate 90 mg/m², cytarabine 225 mg/m²; cycles 5 - 6: if no dose-limiting toxicity occurs in cycles 3 and 4: methotrexate 120 mg/m², cytarabine 300 mg/m²

Level 3

Cycles 1 - 2: methotrexate 90 mg/m², cytarabine 225 mg/m²; cycles 3 - 4: if no dose-limiting toxicity occurs in cycles 1 and 2: methotrexate 120 mg/m², cytarabine 300 mg/m²; cycles 5 - 6: if no dose-limiting toxicity occurs in cycles 3 and 4: methotrexate 150 mg/m², cytarabine 375 mg/m²

Level 4

Cycles 1 - 2: methotrexate 120 mg/m², cytarabine 300 mg/m²; cycles 3 - 6: if no dose-limiting toxicity occurs in cycles 1 and 2: methotrexate 150 mg/m², cytarabine 375 mg/m²

Level 5

Cycles 1 - 6: methotrexate 150 mg/m², cytarabine 375 mg/m²

Phase II

The results of the phase I part of the trial will be summarized and submitted as an interim report to Celgene. Initiation of phase II will require reliable data defining the maximum tolerated dose and demonstration of clinical activity in at least some of the patients treated in phase I.

A total of 20 evaluable patients will be treated at the maximum tolerated dose level. If in phase I three patients were treated at the maximum tolerated dose, another 15 will be added in phase II. If six patients were treated in phase I, another 12 will be included in phase II.

Patients in the phase II part will receive a maximum of 6 treatment cycles. If no dose-limiting toxicity occurs in the first two cycles, the doses of methotrexate and cytarabine may be escalated in cycles 3 and 4, and, in case of no toxicities in cycles 3 and 4, again in cycles 5 and 6. Treatment will be stopped prematurely in case of tumor progression, unacceptable toxicity, intolerance or physician or patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Performance status ECOG 0 - 3
* First or subsequent relapse or refractoriness of a biopsy-proven CD20-positive aggressive B cell lymphoma (excluding mantle cell lymphoma)
* Measurable disease
* Ineligibility or unwillingness to undergo high-dose chemotherapy with autologous stem cell transplantation
* Ability to understand the aim of the study and act accordingly
* Effective contraception
* Signed informed consent

Exclusion Criteria:

* Central nervous system relapse of aggressive lymphoma
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Any condition including the presence of laboratory abnormalities which places the subject at unacceptable risk if he/she were to participate in the study
* Any condition that confounds the ability to interpret data from the study
* Inadequate organ function not related to aggressive lymphoma:

  * neutrophils < 1.0/nl
  * platelets < 75/nl
  * creatinine clearance < 60 ml/min
  * bilirubin ≥ 2,5 mg/dl
  * serum AST/GOT or ALT/GPT ≥ 4 x upper limit of normal
* Active viral hepatitis (HBV, HCV), HIV infection, any other uncontrolled infection
* Pregnancy and nursing period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Two months
  Phase I:
  Dose-limiting toxicity of the combination regimen, determination of the maximum tolerated doses of methotrexate and cytarabine
  Phase II:
  Overall response rate (percentage of complete and partial remissions combined)

SECONDARY OUTCOMES:
Progression-free survival | 1 year

OTHER OUTCOMES:
Relapse rate | 1 year
Event-free survival | 1 year
Disease-free survival | 1 year
Overall survival | 1 year
Toxicity (type, onset, duration) | 1 year
Secondary malignancies | 5 years
Complete remission rate | Six months
Partial remission rate | Six months
Rate of stable disease | Six months
Rate of progressive disease | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Dührsen, MD, Principal Investigator — Klinik für Hämatologie, Universitätsklinikum Essen
Locations (1):
- Klinik für Hämatologie, Universitätsklinikum Essen, Essen, Germany